CLINICAL TRIAL: NCT07166445
Title: Deep Learning for Automated Discrimination Between Stage T1-T2 and T3 Renal Cell Carcinoma on Contrast-Enhanced CT
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUH-2025-RCC-DL-TS001
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Renal Cell; Diagnostic Imaging; Pathology; Deep Learning
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None intervention — this study is retrospective based on the CT images, which dose include any intervention.

SUMMARY:
This study aims to develop and validate a contrast-enhanced CT-based deep-learning model for automatic and accurate preoperative discrimination between T1-T2 and T3 renal cell carcinoma. By quantifying the model's diagnostic performance on an independent test set-using AUC, sensitivity, specificity, positive/negative predictive values, and decision-curve analysis-we will establish a decision-support tool that can be seamlessly integrated into clinical PACS, thereby reducing staging errors, refining surgical planning, and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed renal cell carcinoma on postoperative specimen.
2. Preoperative contrast-enhanced CT performed at our institution with slice thickness ≤ 1 mm and complete DICOM datasets.
3. Postoperative pathologic staging clearly defined as pT1a-T2b or pT3a.
4. CT image quality deemed adequate for analysis.

Exclusion Criteria:

* 1. Pathologic subtype other than RCC. 2. Images with severe artifacts.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery at the Department of Urology, Peking University First Hospital, with postoperative pathological confirmation of renal cell carcinoma (RCC), and who also have complete preoperative contrast-enhanced CT datasets (slice thickness ≤1 mm, lossless DICOM) and definitive pathological staging of pT1a-T2b or pT3a.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance | from 2024 to 2027

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing,, Beijing, China